CLINICAL TRIAL: NCT04914117
Title: Phase 1, First-in-Human, Multicentre, Open-label Study of RC118 for Injection in Patients With Locally Advanced Unresectable/Metastatic Solid Tumours
Brief Title: A Study of RC118 in Patients With Locally Advanced Unresectable/Metastatic Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC118G001
Record Dates: First submitted 2021-05-21; First posted 2021-06-04 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Unresectable Solid Tumor; Metastatic Solid Tumor; Locally Advanced Solid Tumor
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RC118 for injection (Experimental): Part A (Dose Escalation): RC118 will be administered through IV infusion at the various dose levels, including 0.25, 0.5, 1.0, 1.5, 2, 2.5, and 3 mg/kg, 1-12 subjects for each dose level.
  Part B (Dose Confirmation): RC118 will be administered at up to two dose levels, which is equal or lower than MTD/MAD, through IV infusion. Each dose level contains 3-6 subjects.
  Interventions: Drug: RC118 for injection

INTERVENTIONS:
Drug: RC118 for injection — RC118 will be administered intravenously (IV) on Day 1 of every 14-day cycle.

SUMMARY:
This is a Phase 1, First-in-Human, Multicentre, Open-label Study of RC118 for Injection in Patients with Locally Advanced Unresectable/Metastatic Solid Tumours to determine the safety and tolerability of RC118, including the maximum tolerated dose (MTD)/maximum administered dose (MAD), and to define the recommended Phase II dose (RP2D).

DETAILED DESCRIPTION:
This is an open-label, Phase 1, FIH, study consisting of dose-escalation (Part A) and dose confirmation (Part B) in Australia. This trial is to evaluate the safety, tolerability (MTD/MAD), PK, immunogenicity of RC118, and further determine the RP2D. In addition, the preliminary anti-tumour efficacy of RC118 as single agent will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be able to provide documented voluntary informed consent.
2. Male or female patient ≥ 18 years and ≤ 75 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score 0 or 1.
4. The expected survival period exceeds 12 weeks.
5. At least one target lesion that can be measured per Response Evaluation Criteria in Solid Tumours (RECIST) v1.1.
6. Histologically documented, incurable, unresectable locally advanced or metastatic tumours that are intolerable or refractory to standard therapies.
7. Patients agree to provide pre-treatment archived /biopsy tumour samples for retrospective Claudin 18.2 test. Archival tumour tissue should be from the most recent timepoint before entering the trial. In addition, archived samples obtained out of the screening are acceptable if it is discussed and approved by the Investigator and Sponsor in advance. Only when archived samples cannot be obtained, the biopsy will be considered at screening. Fresh tumour biopsies will NOT be considered if significant risk procedures are required with the discretion of Investigator.
8. Adequate bone marrow, liver, and renal function defined as: absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelet ≥ 100 × 109/L, haemoglobin ≥ 90 g/L, serum total bilirubin ≤ 1.5 × upper limit of normal (ULN), ALT, AST or ALP ≤ 2.5 × ULN (≤ 5 × ULN when there is known liver metastasis), serum creatinine ≤ 1.5 × ULN, INR ≤ 1.5 × ULN, APTT ≤ 1.5 × ULN.
9. Willingness to avoid pregnancy or fathering children based on the criteria below:

   * Female patients of childbearing potential and male patients with partners of childbearing potential treated with RC118, must agree to use a highly effective form(s) of contraception during study and within 6 months after the last dose. Those methods include but not limited to combined (oestrogen and progestogen containing) hormonal contraception, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion or vasectomized partner (on the understanding that this is the only one partner during the whole study duration), and sexual abstinence.
   * Females of non-childbearing potential (e.g., surgically sterile with a hysterectomy and/or bilateral oophorectomy or chemically sterile or ≥ 12 months of amenorrhea in the absence of chemotherapy, anti-oestrogens, or ovarian suppression). Those females do not need to undergo pregnancy test.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding.
2. Diagnosed active hepatitis B infection (defined as positive of hepatitis B surface Ag and hepatitis B DNA≥500IU/ml), active hepatitis C infection (defined as presence of hepatitis C RNA), and human immunodeficiency virus infection (defined as positive HIV test) during the screening period.
3. Received vaccines within 4 weeks prior to administration or plan on receiving any vaccine during the study.
4. Subjects with a history of other acquired/congenital immunodeficiency diseases or organ transplantation.
5. Patients have history of targeted therapy of Claudins, or participated in other clinical trials and received investigational product within 4 weeks before the first administration of study drug.
6. Allergic constitution or allergic to known research drug active ingredients or excipient.
7. Patients who are under the treatment of anticoagulant drugs (e.g., warfarin, apixaban, and heparin). Patients using prophylactic doses of heparin (e.g., LMWH) is eligible in the study.
8. Patients undergoing any anti-tumour therapy, including surgery, chemotherapy, radiotherapy and biological therapy, within 4 weeks prior to the first administration of study drug, or palliative radiotherapy for bone/other solitary metastases within 2 weeks prior to the first administration of study drug.
9. Previous adverse reactions resulting from previous anti-tumour therapies, which have not returned to Grade 0 or 1 according to NCI-CTCAE v5.0 (except alopecia) at screening.
10. There are clinical symptoms of fluid in the third space (e.g., large amounts of pleural fluid or ascites) that cannot be controlled by drainage or other therapies.
11. A clinically significant active infection judged by the investigator.
12. Comorbidities that may seriously endanger the patient's safety or affect the completion of the study, such as gastrointestinal bleeding (within 4 weeks prior to the screening period), peptic ulcer, intestinal obstruction, intestinal paralysis, interstitial pneumonia, pulmonary fibrosis, kidney failure, and uncontrolled diabetes.
13. QTc interval > 480 ms in both male and female (based on the mean value of the triplicate screening ECGs); family or personal history of long/short QT syndrome, History of ventricular arrhythmia deemed clinically significant by the investigator, or currently receiving antiarrhythmic drug treatment, or implantation of arrhythmia defibrillation device.
14. History of myocardial infarction within 6 months prior to the screening period, severe or unstable angina pectoris, coronary or peripheral artery bypass grafting, heart failure ≥ 3 (New York Heart Association), or uncontrolled hypertension.
15. Patients with known current alcohol dependence or drug abuse.
16. Patients with a long-term history of systemic steroid therapy. Patients with short-term (≤ 7 days) use and drug withdrawal > 2 weeks are eligible.
17. History or presence of uncontrolled primary brain tumours (e.g., leptomeningeal carcinomatosis) or metastatic brain tumours, unless considered stable by the Investigator and local therapy was completed.
18. History or presence of Grade ≥ 2 peripheral neuropathy.
19. History or presence of uncontrolled mental illness at the discretion of the Investigator, which may place the participant at increased risk of safety/tolerability issues.
20. The patient is, in the opinion of the investigator, expected to be non-compliant with critical trial procedures and is not willing or able to adhere to the trial requirements in the future.
21. Patients who are not appropriate for this clinical trial at the discretion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2023-03-11 (Actual)

PRIMARY OUTCOMES:
MTD/MAD based on number of dose-limiting toxicities (DLTs) | Up to 18 months
  The maximum tolerated dose (MTD)/maximum administered dose (MAD) will be assessed based on the number of patients experiencing DLTs, graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0. If the MTD cannot be reached in this study, the MAD will be recorded.
Determine Recommended Phase 2 Dose (RP2D) | Up to 18 months
  The RP2D may be selected based on the MTD/MAD following consultation with the safety monitoring committee with all available data.
Adverse Events | Up to 18 months
  The adverse events occurring or worsening on or after the first dose of the study drug will be recorded.

SECONDARY OUTCOMES:
Object Response Rate (ORR) | Up to 18 months
  ORR will be determined according to Response Evaluation Criteria in Solid Tumours (RECIST) v1.1. The ORR is defined as the number of patients are either complete response (CR) or partial response (PR), relative to the number of patients belonging to the study of interest.
Progression Free Survival (PFS) | Up to 18 months
  PFS is defined as the time from the date of first administration to the date of the first documentation of progressive disease or death due to any cause, whichever occurs first.
Disease Control Rate (DCR) | Up to 18 months
  DCR is the proportion of patients with disease control.
Duration of response (DOR) | Up to 18 months
  DOR is defined, for patients with response, as the time from first documentation of response (CR or PR) to the date of first documentation of progression of disease or death due to any causes whichever occurs first.
Immunogenicity | Up to 18 months
  Incidence of anti-drug antibody (ADA) against RC118
Maximum Plasma Concentration [Cmax] | Up to 18 months
  Cmax of total antibodies, RC118 and free MMAE
Area under the plasma concentration [AUC] | Up to 18 months
  AUC of total antibodies, RC118 and free MMAE
Tmax | Up to 18 months
  Peak time (Tmax) of total antibodies, RC118 and free MMAE

OTHER OUTCOMES:
CLDN18.2 expression | Up to 18 months
  The expression of CLDN18.2 will be scored semi-quantitatively, based on staining intensity and the percentage of staining in provided archived/biopsy tumor samples

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - Remegen Site #12, Macquarie Park, New South Wales
  - Remegen Site #14, Bedford Park, South Australia
  - Remegen Site #13, Frankston, Victoria
  - Remegen Site #11, Malvern, Victoria

IPD SHARING:
Plan to Share IPD: No